CLINICAL TRIAL: NCT07096349
Title: Multidimensional Assessment of Chronic Pain in Severe Haemophilia A Treated With Monoclonal Antibodies: an Observational Study; an Ambispective Cohort Study
Brief Title: Multidimensional Assessment of Chronic Pain in Severe Haemophilia A
Status: Recruiting | Type: Observational
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, Principal Investigator, Investigación en Hemofilia y Fisioterapia
Other Study IDs: He-MoN
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Hemophilia A Without Inhibitor
Keywords: Hemophilia; Bispecific monoclonal antibodies; Chronic pain; Catastrophising; Self-efficacy; Body image
MeSH Terms: conditions — Hemophilia A; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: Patients with severe haemophilia A from different regions of Spain will be included in the study. Patients who meet the selection criteria will be informed of the characteristics and objectives of the study. They will be provided with an information and informed consent document. After confirming that they do not meet any of the exclusion criteria, the primary and secondary dependent variables and confounding factors will be assessed

SUMMARY:
Introduction: Haemophilia is a congenital coagulopathy characterised by haemarthrosis, mainly in the knees, ankles and elbows. Prophylactic treatment is the most effective therapeutic option for preventing or minimising these bleeds. Bispecific monoclonal antibodies have been shown to be effective in reducing bleeding in patients with haemophilia.

Objectives: To investigate the associations between chronic residual pain and pain catastrophising, perceived self-efficacy regarding the disease and treatment, and body image and perception of visible disability.

Methods. Multicentre cross-sectional cohort studies. 109 patients with severe haemophilia A from different regions of Spain will be included in the study. The primary variable will be chronic residual pain and its functional interference (Brief Pain Inventory-Short Form). Secondary variables will be pain catastrophising (Pain Catastrophising Scale), perceived self-efficacy regarding the disease and treatment (Pain Self-Efficacy Questionnaire), and body image and perception of visible disability (Body Image Scale). Potential confounding variables will include sociodemographic variables (age and educational level), clinical variables (time on monoclonal antibody treatment and number of previous bleeds in the last 12 months) and anthropometric variables (body mass index).

Expected results: It is expected that residual chronic pain will persist in patients with severe haemophilia A treated with monoclonal antibodies and that it will be associated with greater catastrophising, lower self-efficacy and poorer body image, modulating the experience of pain beyond bleeding control.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* With a medical diagnosis of severe haemophilia A (FVIII < 1%).
* No inhibitors to FVIII concentrates at the time of the study.
* At least 3 months of treatment with bispecific monoclonal antibodies.
* Medical diagnosis of haemophilic arthropathy in at least two lower limb joints and ≥5 points on the Haemophilia Joint Health Score.
* Ability to understand and respond to self-administered questionnaires.

Exclusion Criteria:

* Patients diagnosed with severe musculoskeletal or neurological comorbidities causing chronic pain.
* Individuals with neurological or cognitive impairments that prevent them from understanding the questionnaires.
* Patients who have participated in an interventional clinical study in the 6 months prior to the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with haemophilia who meet the selection criteria will be informed of the characteristics of the study and the objectives to be achieved.
  Subjects included in the study will be required to complete a workbook containing a series of questionnaires designed to assess chronic residual pain and pain catastrophising, perceived self-efficacy in relation to the disease and treatment, and body image and perception of visible disability in patients with haemophilia.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2025-10-03 (Estimated); Study Completion 2025-10-26 (Estimated)

PRIMARY OUTCOMES:
Assessment of residual chronic pain and its functional interference at the time of the study. | Screening visit
  Chronic residual pain and its functional interference will be assessed using the Spanish version of the Brief Pain Inventory-Short Form (BPI-SF). This multidimensional self-administered questionnaire explores pain intensity using four items: maximum, minimum, average and current pain, on a scale of 0-10. The degree of interference of pain in daily life is assessed using seven items: mood, activity, work, relationships, sleep, enjoyment of life, and walking, on a scale of 0-10. An average score is calculated for each dimension (intensity and interference). This instrument has shown excellent reliability and validity

SECONDARY OUTCOMES:
Assessment of catastrophising at the time of the study. | Screening visit
  Catastrophising will be assessed using the Spanish version of the Pain Catastrophising Scale (PCS). This self-reported questionnaire consists of 13 items measuring three cognitive dimensions related to pain: rumination, magnification and hopelessness. Each item is scored on a Likert scale from 0 ('never') to 4 ('always'), and the total score ranges from 0 to 52. Higher scores indicate higher levels of catastrophising. This tool has shown excellent internal consistency and test-retest reliability. This scale can predict pain intensity and emotional response in clinical and experimental contexts.
Assessment of perceived self-efficacy for managing chronic pain at the time of the study. | Screening visit
  Perceived self-efficacy for managing chronic pain will be assessed using the Pain Self-Efficacy Questionnaire (PSEQ). This instrument measures the degree to which a person with chronic pain trusts their ability to perform daily activities despite pain. It consists of 10 items, each scored on a 7-point Likert scale ranging from 0 ('not at all confident') to 6 ('completely confident'). The total score ranges from 0 to 60, with higher values indicating greater self-efficacy. The Spanish version of the PSEQ has shown excellent internal consistency and test-retest reliability.
Assessment of body image perception at the time of the study. | Screening visit
  Body image perception will be assessed using the Spanish version of the Body Image Scale (BIS). This instrument, designed for patients after cancer treatment, consists of 10 self-administered items that assess body image distress resulting from this treatment. It uses a 4-point Likert scale (0 = 'not at all' to 3 = 'very much'). The total score ranges from 0 to 30, with higher values indicating greater impairment. The adaptation to Spanish showed excellent internal consistency.

OTHER OUTCOMES:
Assessment of the sociodemographic variable age at the time of the study. | Screening visit
  The sociodemographic variable age will be assessed by calculating the age (in months) from the date of birth to the date of assessment.
Assessment of the sociodemographic variable educational level at the time of the study. | Screening visit
  The sociodemographic variable educational level will be assessed using closed-ended questions (primary education/secondary education/university education/postgraduate education).
Assessment of the clinical variable time with prophylactic treatment with bispecific monoclonal antibodies at the time of the study. | Screening visit
  The clinical variable 'time with prophylactic treatment with bispecific monoclonal antibodies' will be calculated in months (time between the start of treatment with this therapeutic option and the date of evaluation).
Assessment of the variable number of previous joint bleeds in the last 12 months at the time of the study. | Screening visit
  The clinical variable number of previous bleeds in the last 12 months will be calculated based on the number of clinical haemarthrosis. These must meet a series of criteria to be determined as clinical haemarthrosis: inflammation, restricted range of motion, severe pain, functional impairment and the requirement of at least one dose of clotting factor concentrate as rescue treatment.
Assessment of the anthropometric variable body mass index at the time of the study. | Screening visit
  The anthropometric variable body mass index will be calculated using the formula Weight/Height2. To do this, both data will be requested from patients at the time of evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad de Oviedo
Locations (1):
- Universidad de Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No